CLINICAL TRIAL: NCT03669991
Title: Real World Assessment of Effects of Beta-blockers on Patients With Acute Coronary
Brief Title: Real World Assessment of Effects of Beta-blockers on Patients With Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Yi-Da Tang, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 20181082
Record Dates: First submitted 2018-09-03; First posted 2018-09-13 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is aimed to optimized the dose-adjusted regimen of beta-blockers in patients with acute coronary syndrome by investigating therapeutic and curative results of target doses Beta-blockers using the dose-adjusted pathway of beta-blockers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients diagnosed as acute coronary syndromes including acute ST-segment elevation myocardial infarction (STEMI) and non-ST-segment elevated acute coronary syndrome (NSTE-ACS)
* Patients or whose legal representatives signed written informed consent form

Exclusion Criteria:

Patients should been excluded if they meet any of the following exclusion criteria:

* Patients with contraindications to the application of beta blockers, including: 1) cardiogenic shock or heart failure (Killip grade > II level);2) sick sinus syndrome; 3) II degree atrioventricular block;4) unstable decompensation of cardiac failure (pulmonary edema, hypotension or low perfusion); 5) symptomatic hypotension or bradycardia (heart rate<50 beats/min, blood pressure<90/60mmHg); 6) contraindications to beta blockers or allergy to any ingredient of beta blocker; 7) active asthma should be treated by inhalation preparation treatment
* Pregnant or lactating women
* Patients without signed written informed consent
* Patients who was considered by the researcher inappropriate to participate in this study (for example, patients with a higher risk of cardiogenic shock, etc.)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome
Sampling Method: Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2018-08-31 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events (MACCE) | Within 1 year after surgery
  MACCE were defined as a composite of all-cause death, myocardial infarction (MI), unplanned target vessel revascularization (TVR), stent thrombosis (ST) and stroke.

SECONDARY OUTCOMES:
Resting heart rate | Within 1 year after surgery
  The resting heart rate of the body is the number of contractions of the heart that occur in a single minute while the body is at complete rest.
Blood pressure (systolic & diastolic) | Within 1 year after surgery
  Blood pressure (BP) is the pressure of circulating blood on the walls of blood vessels.
Ejection fraction | Within 1 year after surgery
  Ejection fraction (EF) is the volumetric fraction of fluid (usually blood) ejected from a chamber (usually the heart) with each contraction (or heartbeat).
Serum norepinephrine | Within 1 year after surgery
  Norepinephrine is a neurotransmitter that is secreted in response to stress.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Da Tang, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China